CLINICAL TRIAL: NCT00541008
Title: Phase II of Sunitinib (SUTENT®) in First Line for Patients With Locally Advanced or Metastatic Papillary Renal Cell Carcinoma - SUPAP
Brief Title: Sunitinib as First-Line Therapy in Treating Patients With Locally Advanced Metastatic Papillary Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000569863; FRE-FNCLCC-GEP-03-0603; EU-20761; EUDRACT-2006-003339-62; PFIZER-FRE-FNCLCC-GEP-03-0603
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Kidney Cancer
Keywords: type 1 papillary renal cell carcinoma; type 2 papillary renal cell carcinoma; stage IV renal cell cancer; stage III renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: sunitinib malate

SUMMARY:
RATIONALE: Sunitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works as first-line therapy in treating patients with locally advanced or metastatic papillary renal cell (kidney) cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the objective tumor response rate in patients with locally advanced or metastatic papillary renal cell carcinoma treated with sunitinib malate.

Secondary

* To evaluate the safety of this drug in these patients.
* To determine time-to-event variables of overall survival, time to disease progression, time to response, and duration of response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate once a day on days 1-28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 28 days and then periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of papillary renal cell carcinoma

  * Locally advanced or metastatic disease
  * Type I or type II disease
* Progressive disease
* Measurable disease defined by RECIST criteria as at least 1 lesion at least 2 cm in length by conventional CT scan techniques or at least 1 cm by spiral CT scan
* No brain metastases including treated and nonprogressive metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8 g/dL
* Total bilirubin ≤ 3 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Serum creatinine < 1.5 times ULN
* INR ≤ 1.7 or PT ≤ 6 seconds over ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Patients must be affiliated to a Social Security System
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion criteria:

* NCI CTC grade 3 hemorrhage within 4 weeks prior to start of study treatment
* Diagnosis of any second malignancy within the past 3 years except for basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma of the cervix that has been adequately treated with no evidence of recurrent disease within the past 12 months
* Spinal cord compression, carcinomatous meningitis, or leptomeningeal disease
* Any of the following within the past 12 months prior to study drug administration:

  * Severe/unstable angina
  * Myocardial infarction
  * Coronary artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident including transient ischemic attack
  * Pulmonary embolism
* Any of the following conditions:

  * Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2
  * Atrial fibrillation of any grade
  * Prolongation of the QTc interval to > 450 msec for males or > 470 msec for females
* Hypertension that cannot be controlled by medications
* Inability to swallow oral medications or presence of active inflammatory bowel disease, partial or complete bowel obstruction, or chronic diarrhea
* Known HIV or AIDS infection
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration
* Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and the follow-up schedule
* Patients deprived of liberty or placed under the authority of a tutor

PRIOR CONCURRENT THERAPY:

* Recovered from all toxic effects of any prior local treatment to CTCAE version 3.0 grade ≤ 1
* At least 4 weeks since prior radiotherapy

  * At least 1 week since prior radiotherapy to < 10% of the whole body allowed provided side effects are < grade 2 and there is at least one site for evaluation
* More than 2 weeks since prior and no concurrent anticoagulant agents or therapeutic doses of warfarin

  * Low-dose warfarin (up to 2 mg/day) for deep vein thrombosis prophylaxis allowed
  * Low molecular weight heparin allowed
* No prior specific medical systemic therapy (i.e., first-line therapy)
* No prior sunitinib malate
* No prior investigational agents
* No concurrent treatment on another therapeutic clinical trial

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-09-05 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate

SECONDARY OUTCOMES:
Safety
Overall survival
Time to disease progression
Time to response
Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Alain Ravaud, MD, PhD — Hopital Saint Andre
Locations (22):
- France (22):
  - Centre Paul Papin, Angers
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Saint Andre, Bordeaux
  - C.H.U. de Brest, Brest
  - Centre Regional Francois Baclesse, Caen
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Saint Michel, Paris
  - Institut Jean Godinot, Reims
  - Hopital Foch, Suresnes
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Cabarrou B, Boher JM, Bogart E, Tresch-Bruneel E, Penel N, Ravaud A, Escudier B, Mahier Ait-Oukhatar C, Delord JP, Roche H, Filleron T. How to report toxicity associated with targeted therapies? Ann Oncol. 2016 Aug;27(8):1633-8. doi: 10.1093/annonc/mdw218. Epub 2016 May 23. PMID 27217543
- [Derived] Ravaud A, Oudard S, De Fromont M, Chevreau C, Gravis G, Zanetta S, Theodore C, Jimenez M, Sevin E, Laguerre B, Rolland F, Ouali M, Culine S, Escudier B. First-line treatment with sunitinib for type 1 and type 2 locally advanced or metastatic papillary renal cell carcinoma: a phase II study (SUPAP) by the French Genitourinary Group (GETUG)dagger. Ann Oncol. 2015 Jun;26(6):1123-1128. doi: 10.1093/annonc/mdv149. Epub 2015 Mar 23. PMID 25802238